CLINICAL TRIAL: NCT02898675
Title: Investigation of the Contributions of Platelet Rich Fibrin Combined With Open Flap Debridement on Periodontal Healing
Brief Title: Advantages of Autologous Platelet-Rich Fibrin Membrane on Growth Factor Levels and Periodontal Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Taner ARABACI, Clinical Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAP-2011300
Record Dates: First submitted 2016-08-24; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet Rich Fibrine (Experimental): Platelet Rich Fibrine was applied with open flap debridement in test group.
  Interventions: Device: Platelet rich fibrine
- Open Flap Debridement (Active Comparator): Platelet Rich Fibrin was not applied to control groups. Only open flap debridement was applied to control groups.
  Interventions: Device: Open Flap Debridement

INTERVENTIONS:
Device: Platelet rich fibrine — Platelet rich fibrin increases the growth factors. So it was applied for treatment of periodontal bone loss.
  Arms: Platelet Rich Fibrine
Device: Open Flap Debridement — Only open flap debridement treatment the bone loss limitedly
  Arms: Open Flap Debridement

SUMMARY:
Platelet rich fibrin is a second generation platelet concentration which contains various growth factors. The aim of this study is to evaluate the clinical and biochemical efficacy of PRF in subjects of chronic periodontitis in the operation of conventional periodontal flap.

DETAILED DESCRIPTION:
PRF was developed in 2001 by Choukroun in France, it was the second generation fibrin adhesive, and was used to accelerate the soft and hard tissue healing. Many studies have shown beneficial effects of PRF on osteoconductive filler material in sinus lift operations, treatment of periodontal sulcus defect and treatment of furcation defects. Also PRF contains many growth factors. PRF accelerates periodontal regeneration through the gradually excreted growth factors and contributes to the bone regeneration. In this study, the investigators evaluated the effect of PRF on growth factors and its contribution to periodontal regeneration in subjects with chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CP who had pocket depth ≤ 5 mm and at least two area (grouped as Control and PRF) with horizontal bone loss after initial treatment

Exclusion Criteria:

* The subjects excluded in the study had history of systemic disease, were smokers, had allergy to any drug, had need for prophylaxis of antibiotic and had taken antibiotics at least 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Level of Growth Factor | 6 weeks
  Change from baseline growth factors levels of GCF at 6 weeks were measured by periopaper

SECONDARY OUTCOMES:
Alteration of Clinical Attachment Level | 9 month
  Change from baseline Clinical Attachment Levels at 9 months were measured with periodontal probe.
Alteration of Periodontal Pocket Depth | 9 month
  Change from baseline Pocket Depth at 9 months were measured with periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Yasin ÇİÇEK, Study Chair — Adiyaman University

REFERENCES:
- [Background] Pradeep AR, Shetty SK, Garg G, Pai S. Clinical effectiveness of autologous platelet-rich plasma and Peptide-enhanced bone graft in the treatment of intrabony defects. J Periodontol. 2009 Jan;80(1):62-71. doi: 10.1902/jop.2009.080214. PMID 19228091
- [Derived] Arabaci T, Kose O, Albayrak M, Cicek Y, Kizildag A. Advantages of Autologous Platelet-Rich Fibrin Membrane on Gingival Crevicular Fluid Growth Factor Levels and Periodontal Healing: A Randomized Split-Mouth Clinical Study. J Periodontol. 2017 Aug;88(8):771-777. doi: 10.1902/jop.2017.160485. Epub 2017 Apr 28. PMID 28452623